CLINICAL TRIAL: NCT01458626
Title: A Double-blind, Active-controlled, Randomized Study Comparing Mirtazapine Combined With Paroxetine or Paroxetine Monotherapy in Patients With Major Depressive Patients Without Early Improvement in the First 2 Weeks
Brief Title: Effectiveness Study of Mirtazapine Combined With Paroxetine in Major Depressive Patients Without Early Improvement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Gang Wang, MD, Head of Depression Center, Capital Medical University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: MISP # 39888
Record Dates: First submitted 2011-08-09; First posted 2011-10-25 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Major Depression
Keywords: mirtazapine; paroxetine; major depression; early improvement
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Mirtazapine; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Add-on therapy (Active Comparator): mirtazapine 30mg QD and paroxetine 20mg QD
  Interventions: Drug: mirtazapine; Drug: paroxetine 20mg QD
- mirtazapine monotherapy (Active Comparator): mirtazapine 30mg QD
  Interventions: Drug: mirtazapine
- paroxetine monotherapy (Active Comparator): paroxetine 20mg QD
  Interventions: Drug: paroxetine 20mg QD

INTERVENTIONS:
Drug: mirtazapine — mirtazapine 30mg QD
  Other Names: Remeron
  Arms: Add-on therapy; mirtazapine monotherapy
Drug: paroxetine 20mg QD — paroxetine 20mg QD
  Other Names: Seroxat
  Arms: Add-on therapy; paroxetine monotherapy

SUMMARY:
Although treatment guidelines manifest that antidepressant response usually appear with a delay of several weeks and suggest that treatment should be changed if a partial response has not occurred after 4~6 week, these beliefs are no longer held by experts, and a new concept is raised that the first 2 weeks of treatment may be a useful strategy for improving the management of depression. New evidence indicates that early treatment response can be predicted with high sensitivity after 2 weeks of treatment in patients with major depressive disorder (MDD).

Early improvement not only predicted response or remission, but also that lack of improvement was associated with little chance of response if the treatment strategy remained unchanged. The criterion of a 20% score reduction has been chosen as an early indicator of improvement because it can be reliably measured in clinical trials and translates into a clinically relevant change in the severity of depressive symptoms.

Antidepressants that enhance both serotonergic and noradrenergic neurotransmission may be more effective than selective serotonin reuptake inhibitors (SSRIs) for acute-phase therapy of major depressive disorder. As a noradrenergic and specific serotonergic antidepressant, the antidepressive mechanism of mirtazapine is quite superior to SSRI and in particular has been suggested to have a faster onset of action than SSRIs in MDD patients.

The aim of this study is to provide physicians with further information regarding early improvement and the effectiveness of mirtazapine combined with a SSRI antidepressant therapy in nonresponders.

DETAILED DESCRIPTION:
Mirtazapine has significant advantages in response and remission rates compared with various SSRIs in double-blind treatment. Mirtazapine combined with SSRIs or venlafaxine was also found to be one of the more effective and successful strategy for nonresponders in MDD. The investigators hypothesized that mirtazapine as adjunctive treatment to paroxetine can boost the onset time and also can improve the antidepression action of SSRIs in patients without early improvement.

The aim of this study is to provide physicians with further information regarding early improvement and mirtazapine combined with a SSRI antidepressant therapy in nonresponders, by providing a comparison of depressive symptoms outcomes associated with adjunctive mirtazapine or mono- paroxetine in MDD patients who have previously been treated with paroxetine for 2 weeks and who have not attained improvement. Paroxetine has been chosen as a comparator because it is a widely-used and relatively well-tolerated SSRI antidepressant.

The study is designed as a multi-center, randomized, double-blind, active-controlled trial in subjects with MDD.

Patients will be male or female, 18 to 60 years of age, inclusive, outpatient or inpatient status, with diagnosis of major depressive episode (single or recurrent) by DSM-IV. The patients should also have HAMD-17 total score ≥ 20,a HAMD-17 Item 1(depressed mood) score ≥ 2 at enrollment in open-label preliminary phase.

It will consist of 2 phases. An open-label preliminary phase lasts for 2 weeks, during which paroxetine is titrated up to 20mg/day (Day 5). At Week 2, patients will be evaluated by HAMD-17. The patients who have achieved early improvement (the decrease of HAMD-17 total score ≥ 20%) will be discontinued. The patients who have not achieved early improvement (the decrease of HAMD-17 total score < 20%), will be randomized into three treatment arms [1.Mirtazapine (30mg/d); 2.Paroxetine (20mg/d); 3.Mirtazapine (30mg/d) +Paroxetine(20mg/d)]. In double-blind treatment phase (consist of 6 weeks), patients will be evaluated at Week 3, 4, 6 and 8.

Primary efficacy measure will be assessed based on the decrease of HAMD-17 from randomization (Week 2) to endpoint (Week 8). CGI-I and CGI-S will be used as secondary efficacy measures throughout this phase.

The safety in this study will be assessed by adverse event reporting, clinical laboratory measurements and physical examinations.

Up to 540 patients will enter into Open-label Phase in order to yield approximately 200 evaluable patients in Randomization Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Has given written informed consent.
2. Male or female outpatients aged at least 18 years and not more than 60 years.
3. Has a diagnosis of major depressive disorder by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria.
4. HAMD-17 ≥ 20 and HAMD-17 Item 1(depressed mood) score ≥2 at enrolment in open-label preliminary phase.

Exclusion Criteria:

1. Currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug.
2. Current Axis I primary psychiatric diagnosis other than major depressive disorder.
3. Organic mental disease, including mental retardation.
4. History of clinically significant disease, including any cardiovascular, hepatic, renal, respiratory, hematologic, endocrinologic, or neurologic disease, or clinically significant laboratory abnormality that is not stabilized or is anticipated to require treatment during the study.
5. Subjects receiving an investigational agent (including different formulation and generic agents of investigational drug) in the previous 3 months prior to screening.
6. Women in pregnancy or lactation, or female of child bearing potential without appropriate birth control measures.
7. Use of antipsychotics or mood stabilizers within 5 days prior to screening.
8. Has received depot antipsychotic medication within one cycle prior to screening.
9. Known allergy or lack of response to mirtazapine.
10. Has received ECT or MECT within 3 months prior to screening.
11. Significant risk of suicidal and/or self-harm behaviors.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 525 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2016-08-24 (Actual)

PRIMARY OUTCOMES:
Symptoms Improvement by HAMD-17 | From randomization (Week 2) to endpoint(Week 8)
  Change of 17-item Hamilton Depression Scale (HAMD-17) total score

SECONDARY OUTCOMES:
Self-reported improvement by QIDS-SR | From randomization (Week 2) to endpoint(Week 8)
  Change of Quick Inventory of Depressive Symptomatology-self report (QIDS-SR) total score
Remission rate by HAMD-17 | From randomization (Week 2) to endpoint(Week 8)
  The proportion of subjects at endpoint with HAMD-17 total score ≤7
Remission rate by QIDS-SR | From randomization (Week 2) to endpoint(Week 8)
  The proportion of subjects at endpoint with QIDS-SR total score ≤5
Response rate HAMD-17 | From randomization (Week 2) to endpoint(Week 8)
  The proportion of subjects at endpoint with the reduction of HAMD-17 total score >=50%
Response rate by QIDS-SR | From randomization (Week 2) to endpoint(Week 8)
  The proportion of subjects at endpoint with the reduction of QIDS-SR total score >=50%
Clinical Global Impression-improvement | Endpoint(Week 8)
  The proportion of subjects at endpoint with CGI-I as "much improved" or "very much improved"
Clinical Global Impression- severity | From randomization (Week 2) to endpoint(Week 8)
  Change of CGI-S total score
Safety outcome 1 | From enrollment to endpoint (Week 8)
  The incidence and nature of overall adverse events
Safety outcome 2 | From enrollment to endpoint (Week 8)
  The incidence and nature of drug-related adverse events
Drop-off rate due to adverse events | From randomization (Week 2) to endpoint(Week 8)
  The number of subject withdrawal due to adverse events during double-blind phase

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, M.D., Ph.D, Principal Investigator — Beijing Anding Hospital, Capital Medical University
Locations (1):
- Beijing Anding Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhou J, Liu S, Mayes TL, Feng Y, Fang M, Xiao L, Wang G. The network analysis of depressive symptoms before and after two weeks of antidepressant treatment. J Affect Disord. 2022 Feb 15;299:126-134. doi: 10.1016/j.jad.2021.11.059. Epub 2021 Nov 24. PMID 34838606